CLINICAL TRIAL: NCT01560611
Title: The Somatic-to-cerebral Oxygen Saturation Gradient as a Non-invasive Index of Anaerobic Threshold in High-risk Cardiac Surgical Patient
Brief Title: A New Non-invasive Marker to Detect Silent Hypoxia in Patients Undergoing Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5162
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Cardiac Surgical Procedures; High-risk Surgical Patient; Anaerobic Threshold
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- High-risk cardiac surgery patient
  Interventions: Device: Near infrared spectroscopy

INTERVENTIONS:
Device: Near infrared spectroscopy

SUMMARY:
In patients undergoing cardiac surgery under cardiopulmonary bypass, some organs like brain and heart are preserved while others (skin, gut and skeletal muscle) are being underperfused. This phenomenon is related to silent peripheral vasoconstriction that is not clinically available but threatens end-organ perfusion and carries the risk of multi-organ failure. By measuring non-invasively the somatic-to-cerebral oxygen saturation gradient, the present study aims at detecting silent peroperative hypoperfusion episodes. The investigators hypothesize that gradient, measured during the surgical procedure, will predict the occurrence of anaerobic metabolism, ascertained by an elevation of blood lactate concentration, measured in intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yo
* Cardiac surgical procedure under cardiopulmonary bypass
* High-risk surgical patient fulfilling one of the following items:

  * Euroscore >= 6
  * Ejection fraction < 40%
  * Creatinine clearance < 40mL/min
  * Pulmonary arterial pressure > 45mmHg
* Signed informed consent
* Social security affiliation

Exclusion Criteria:

* Emergency situation
* Patient on ECMO
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgical procedures under cardiopulmonary bypass in Strasbourg University Hospital
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-03

CONTACTS AND LOCATIONS:
Overall Officials: Julien POTTECHER, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Pôle d'anesthésie réanimation - Nouvel Hôpital Civil, Strasbourg, France